CLINICAL TRIAL: NCT04845750
Title: The RODEO Micro Mapping Catheter in Cryoablation Procedures - A Feasibility Study
Brief Title: The RODEO Micro Mapping Catheter in Cryoablation Procedures
Acronym: RODEO-MaPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: afreeze GmbH (Other)
Collaborators: Competence Center for Medical Devices GmbH (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RODEO-MaPS
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases
Keywords: Atrial Fibrillation; Paroxysmal Atrial Fibrillation; Persistent Atrial Fibrillation; Cryoablation; Cryosurgery; Mapping Catheter
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Cardiovascular Diseases; Heart Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rodeo Micro Mapping Catheter (Experimental): Determination of pulmonary vein isoation during cryoablation procedure
  Interventions: Device: Rodeo Micro Mapping Catheter

INTERVENTIONS:
Device: Rodeo Micro Mapping Catheter — The Rodeo Micro Mapping Catheter is used during cryoablation of atrial fibrillation patients for determination of pulmonary vein isolation

SUMMARY:
This clinical investigation evaluates the feasibility of the Rodeo Micro Mapping Catheter in combination with cryoablation ssystem (sclerotherapy of muscle tissue of the heart by freezing) in patients with atrial fibrillation (permanent atrial fibrillation excepted).

Further aims of this study are the evaluation of safety of the device and average procedure and fluoroscopy times.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and legal capacity.
* Atrial fibrillation, diagnosed in accordance with the guidelines of the ESC (version 2016) - permanent AF excluded.
* Patient planned for a pulmonary vein isolation catheter ablation procedure using cryoenergy and suitable for treatment according to the respective instructions for use (IFU).
* Signed and dated informed consent documented by the patient, indicating that the patient has been informed of all the pertinent aspects of the trial prior to study enrolment (patient has received a copy of the ICF).

Exclusion Criteria:

* Indication that the vascular system is not accessible through the left or right groin.
* Indication that a transseptal puncture cannot be performed.
* Any previous ablation or surgery due to AF.
* Important comorbidities such as cardiovascular events within six months of enrolment or high-risk surgical patients.
* Left atrial diameter > 50 mm in the short axis.
* Advanced structural heart disease including

  * moderate-to-severe valvular stenosis or regurgitation,
  * previous valve replacement or valve repair,
  * congenital heart disease,
  * left ventricular ejection fraction < 45% during sinus rhythm,
  * congestive heart failure NYHA III or IV,
  * coronary artery bypass graft surgery within the last 3 months.
* Permanent pacemaker.
* Pregnant women at the time of the cryoablation procedure.
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the Informed Consent Form.
* Participation in interventional trials for cardiovascular devices or drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the Rodeo Micro Mapping Catheter | 1-3 hours
  Percentage of pulmonary veins with diagnostically conclusive signals measured with the RODEO Micro Mapping Catheter.
Positioning of the Rodeo Micro Mapping Catheter | 1-3 hours
  Percentage of pulmonary veins where positioning of the cryoablation catheter with the Rodeo Micro Mapping Catheter as guidewire was possible

SECONDARY OUTCOMES:
Safety of the Rodeo Micro Mapping Catheter. | 1-3 day follow-up period
  Percentage of adverse events related to the Rodeo Micro Mapping Catheter
Efficacy of the Rodeo Micro Mapping Catheter | 1-3 hours
  Percentage of successfully isolated pulmonary veins
Real-time pulmonary vein isolation | 1-3 hours
  Time from beginning of the freeze to conduction blockade (time to effect)
Procedural safety | 1-3 hours
  Procedure-related adverse events
Total procedure time | 1-3 hours
  Total procedure time defined from introduction of the transseptal sheath until removal of the transseptal sheath
Cryoablation catheter procedure time | 1-3 hours
  Cryoablation catheter procedure time defined from introduction of the cryoablation catheter into the left atrium until removal of the cryoablation catheter from the left atrium after termination of the last cryo-application
Total fluoroscopy time and dose | 1-3 hours
  Total fluoroscopy time and dose defined from introduction of the transseptal sheath until removal of the transseptal sheath
Cryoablation catheter fluoroscopy time and dose | 1-3 hours
  Cryoablation catheter fluoroscopy time and dose defined from introduction of the cryoablation catheter into the left atrium until removal of the cryoablation catheter from the left atrium after termination of the last cryo-application

CONTACTS AND LOCATIONS:
Overall Officials: Florian Hintringer, MD, Principal Investigator — Medizinische Universität Innsbruck
Locations (2):
- Medizinische Universität Innsbruck, Innsbruck, Tyrol, Austria
- Marienhaus Klinikum St. Elisabeth Neuwied, Neuwied, Rhineland-Palatinate, Germany